CLINICAL TRIAL: NCT07385352
Title: Comparative Evaluation of Caudal Dexmedetomidine and Caudal Ketamine as Adjuvants to Isobaric Bupivacaine for Postoperative Analgesia in Children Undergoing Surgery for Developmental Dysplasia of the Hip
Brief Title: Caudal Dexmedetomidine vs Ketamine for Postoperative Analgesia in Pediatric DDH Surgery
Acronym: CDK-DDH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Abdelmonem Ahmed Mahmoud, Resident of Anesthesiology, Assiut University Hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-2026-201643
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Developmental Dysplasia of the Hip
Keywords: Caudal block Dexmedetomidine Ketamine Pediatric analgesia Bupivacaine Postoperative pain Hip surgery DDH
MeSH Terms: conditions — Developmental Dysplasia of the Hip | interventions — Dexmedetomidine; Ketamine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Children are randomized to receive either Dexmedetomidine or Ketamine as adjuvant to caudal Bupivacaine for postoperative analgesia following developmental dysplasia of the hip (DDH) surgery.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double-blind study: neither the patient, the anesthesiologist administering the block, nor the assessor recording pain scores will be aware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Experimental): Children receiving caudal Isobaric Bupivacaine 0.25% (1 ml/kg) with Dexmedetomidine 1 µg/kg for postoperative analgesia.
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacaine
- Ketamine Group (Experimental): Children receiving caudal Isobaric Bupivacaine 0.25% (1 ml/kg) with Ketamine 0.5 mg/kg for postoperative analgesia.
  Interventions: Drug: Ketamine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 1 µg/kg added to caudal Bupivacaine.
  Arms: Dexmedetomidine Group
Drug: Ketamine — Ketamine 0.5 mg/kg added to caudal Bupivacaine.
  Arms: Ketamine Group
Drug: Bupivacaine — Isobaric Bupivacaine 0.25% 1 ml/kg used for caudal block in both groups.

SUMMARY:
This study compares two medicines, Dexmedetomidine and Ketamine, added to caudal Bupivacaine to control pain after hip surgery in children. We will check how well each medicine reduces pain, how long the pain relief lasts, and if children need extra pain medicine. The goal is to find the safest and most effective option for postoperative pain relief in children undergoing hip surgery.

DETAILED DESCRIPTION:
Background:

Postoperative pain control is a major concern in pediatric patients undergoing surgery for developmental dysplasia of the hip (DDH). Caudal epidural block with Isobaric Bupivacaine is a common technique, but its duration of analgesia is limited. Adjuvants such as Dexmedetomidine and Ketamine may prolong analgesia and improve postoperative comfort.

Objective:

To compare the efficacy and safety of caudal Dexmedetomidine versus caudal Ketamine as adjuvants to Isobaric Bupivacaine for postoperative analgesia in children undergoing DDH surgery.

Study Design:

Randomized, double-blind, parallel-group clinical trial Participants: Pediatric patients scheduled for DDH corrective surgery

Interventions:

Group A: Caudal Bupivacaine + Dexmedetomidine Group B: Caudal Bupivacaine + Ketamine

Outcomes:

Primary: Postoperative pain scores using FLACC scale Secondary: Duration of analgesia, need for rescue analgesia, hemodynamic stability, and adverse effects

Significance:

This study aims to provide evidence for the most effective and safe adjuvant for pediatric caudal analgesia, reducing opioid use and improving postoperative comfort and recovery in children undergoing hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 6 years undergoing surgery for developmental dysplasia of the hip
* ASA physical status I or II
* Parental or guardian informed consent obtained

Exclusion Criteria:

* Known allergy to local anesthetics, Dexmedetomidine, or Ketamine
* Coagulopathy or bleeding disorders
* Infection at the site of caudal injection
* Neurological disorders
* Severe systemic disease
* Refusal of parental consent

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score (FLACC) | First 24 hours post-surgery
  Pain will be assessed using the FLACC scale (Face, Legs, Activity, Cry, Consolability) at regular intervals (every 2-4 hours) during the first 24 hours after surgery to evaluate the effectiveness of caudal analgesia in children receiving Dexmedetomidine or Ketamine as adjuvants to Bupivacaine.

SECONDARY OUTCOMES:
Hemodynamic Stability | Intraoperative and first 24 hours post-surgery
  Monitoring blood pressure and heart rate intraoperatively and postoperatively to assess safety of caudal adjuvants.
Duration of Analgesia | From caudal block to first request for rescue analgesia
  Time from caudal block administration to first request for rescue analgesia, measured in hours, to compare the prolongation of analgesia between Dexmedetomidine and Ketamine groups.
Adverse Effects | First 24 hours post-surgery
  Recording any side effects related to caudal adjuvants, including bradycardia, hypotension, nausea, vomiting, and sedation, during the first 24 hours.
Rescue Analgesia Requirement | First 24 hours post-surgery
  Number of patients requiring additional analgesia within the first 24 hours post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Esraa Abdelmonem, MSc, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this study will be shared upon reasonable request from qualified researchers. Data will include demographic data, intraoperative and postoperative analgesic parameters, pain scores, and adverse events, after removal of all personal identifiers.
Time Frame: Beginning 6 months following publication and ending 5 years after publication.
Access Criteria: Access will be provided to researchers with a methodologically sound proposal, after approval by the principal investigator and institutional ethics committee. Data will be shared for purposes of achieving the aims of the approved proposal. A data access agreement will be required.

REFERENCES:
- [Background] Yoon JH, Park J, Conde J, Wakamiya M, Prakash L, Prakash S. Rev1 promotes replication through UV lesions in conjunction with DNA polymerases eta, iota, and kappa but not DNA polymerase zeta. Genes Dev. 2015 Dec 15;29(24):2588-602. doi: 10.1101/gad.272229.115. PMID 26680302
- [Background] Tait AR, Burke C, Voepel-Lewis T, Chiravuri D, Wagner D, Malviya S. Glycopyrrolate does not reduce the incidence of perioperative adverse events in children with upper respiratory tract infections. Anesth Analg. 2007 Feb;104(2):265-70. doi: 10.1213/01.ane.0000243333.96141.40. PMID 17242078
- [Background] Zink W, Graf BM. Local anesthetic myotoxicity. Reg Anesth Pain Med. 2004 Jul-Aug;29(4):333-40. doi: 10.1016/j.rapm.2004.02.008. PMID 15305253
- [Background] Beckie TM, Beckstead JW, Groer MW. The influence of cardiac rehabilitation on inflammation and metabolic syndrome in women with coronary heart disease. J Cardiovasc Nurs. 2010 Jan-Feb;25(1):52-60. doi: 10.1097/JCN.0b013e3181b7e500. PMID 19935427
- [Background] Mokta KK, Kanga AK, Kaushal RK. Neonatal listeriosis: a case report from sub-Himalayas. Indian J Med Microbiol. 2010 Oct-Dec;28(4):385-7. doi: 10.4103/0255-0857.71824. PMID 20966576